CLINICAL TRIAL: NCT03075553
Title: Phase 2 Single-Arm, Open-Label Study of Nivolumab in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma (PTCL)
Brief Title: Nivolumab in Treating Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to poor response
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1681; NCI-2017-00307 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1681 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2017-03-01; First posted 2017-03-09 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2019-05

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm; Hepatosplenic T-Cell Lymphoma; HTLV-1 Infection; NK-Cell Lymphoma, Unclassifiable; Primary Systemic Anaplastic Large Cell Lymphoma, ALK-Negative; Recurrent Adult T-Cell Leukemia/Lymphoma; Recurrent Anaplastic Large Cell Lymphoma; Recurrent Angioimmunoblastic T-cell Lymphoma; Recurrent Enteropathy-Associated T-Cell Lymphoma; Recurrent Mycosis Fungoides; Refractory Adult T-Cell Leukemia/Lymphoma; Refractory Anaplastic Large Cell Lymphoma; Refractory Angioimmunoblastic T-cell Lymphoma; Refractory Enteropathy-Associated T-Cell Lymphoma; Refractory Mycosis Fungoides; Refractory Nasal Type Extranodal NK/T-Cell Lymphoma; Refractory Peripheral T-Cell Lymphoma, Not Otherwise Specified
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm; HTLV-I Infections; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma; Mycosis Fungoides; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1. Treatment repeats every 14 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease, complete response, or partial response receive nivolumab IV over 60 minutes on day 1 of course 9. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab works in treating patients with peripheral T-cell lymphoma that has come back after a period of improvement or that does not respond to treatment. Monoclonal antibodies, such as nivolumab, may block cancer growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical benefit of nivolumab in T-cell lymphomas, as measured by objective response rate (ORR) within 12 cycles according to the Lugano Classification Response Criteria (2014).

SECONDARY OBJECTIVES:

I. To assess safety and tolerability of the regimen in this patient population. II. To assess progression-free survival (PFS). III. To assess duration of response (DOR). IV. To assess overall survival (OS).

TERTIARY OBJECTIVES:

I. To evaluate T-cell/cytokine profile in the peripheral blood - peripheral blood specimens will be used to assess T-cell activation and cytokine up regulation as measures of treatment effect.

II. To evaluate intratumoral biomarkers- intratumoral cell populations and distribution, genetic variability, mutational burden and T-cell activation will be evaluated to identify potential biomarkers that correlate with response to therapy.

III. To assess the potential association between PD-L1/PD-1/PD-L2 expression on tumor and T-cells and/or PD-L1 soluble levels in plasma with clinical efficacy of PD-1 blockade.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 60 minutes on day 1. Treatment repeats every 14 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease, complete response, or partial response receive nivolumab IV over 60 minutes on day 1 of course 9. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 35 days, 100-120 days, 230-250 days, and 330-390 days.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory T-cell lymphoma (TCL) biopsy-proven =< 6 months prior to registration, including the following subtypes:

  * Peripheral T-cell lymphoma, not otherwise specified
  * Anaplastic large cell lymphoma, anaplastic lymphoma kinase (ALK) negative, primary systemic type
  * Angioimmunoblastic T-cell lymphoma
  * Extranodal natural killer (NK)/T-cell lymphoma, nasal type
  * Adult T-cell lymphoma/leukemia (human T-lymphotropic virus 1 [HTLV1]+)
  * Blastic NK-cell lymphoma
  * Enteropathy-associated T-cell lymphoma
  * Hepatosplenic gamma delta T-cell lymphoma
  * Transformed mycosis fungoides
  * T/NK-cell lymphoma, unclassifiable
* Measurable disease: subjects must have at least one lesion that is > 15mm (1.5 cm) in the longest diameter on cross-sectional imaging and measureable in two perpendicular dimensions per computed tomography (spiral CT) or magnetic resonance imaging (MRI)
* After failure of allogeneic stem cell transplant (ASCT) or after failure of frontline therapy in subjects who declined or are not ASCT candidates
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* White blood cell (WBC) >= 3000/mm^3
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless elevation due to Gilbert's Syndrome
* Aspartate transaminase (AST) =< 2.5 x ULN
* Creatinine =< 2.0 mg/dL
* Calculated creatinine clearance must be >= 45 ml/min using the Cockcroft-Gault formula
* Negative serum or urine pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only Note: Persons of child-bearing potential (POCBP) must use appropriate method(s) of contraception; POCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug; men who are sexually active with POCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with POCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; persons who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception; should a person become pregnant or suspect being pregnant while participating in this study, the person should inform the treating physician immediately
* Provide written informed consent
* Willing to return to enrolling institution for follow-up during the Active Monitoring phase of the study
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* All primary cutaneous T-cell lymphomas
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Active, known or suspected autoimmune disease Note: subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment
* Use of systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications < 14 days of registration Note: inhaled or topical steroids are permitted; > 10 mg daily prednisone equivalents are permitted only in adrenal insufficiency in the absence of active autoimmune disease
* Prohibited treatments and or therapies

  * Autologous stem cell transplant (ASCT) =< 12 weeks prior to first dose of the study drug
  * Prior treatments (window prior to registration):

    * Chemotherapy =< 2 weeks
    * Nitrosureas =< 6 weeks
    * Therapeutic anticancer antibodies =< 4 weeks
    * Radio- or toxin immunoconjugates =< 10 weeks
    * Radiation therapy =< 3 weeks
    * Or major surgery =< 2 weeks
  * Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways

    * Prior allogeneic stem cell transplant (SCT)
    * Chest radiation =< 24 weeks prior to registration
* Immunocompromised patients, patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) and currently receiving antiretroviral therapy, active hepatitis B virus surface antigen (HBV sAg+), active hepatitis C (if Ab+ then PCR+) indicating acute or chronic infection
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Active central nervous system (CNS) involvement or leptomeningeal involvement
* History of pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ansell, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bennani NN, Kim HJ, Pederson LD, Atherton PJ, Micallef IN, Thanarajasingam G, Nowakowski GS, Witzig T, Feldman AL, Ansell SM. Nivolumab in patients with relapsed or refractory peripheral T-cell lymphoma: modest activity and cases of hyperprogression. J Immunother Cancer. 2022 Jun;10(6):e004984. doi: 10.1136/jitc-2022-004984. PMID 35750419

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nivolumab): Patients receive 240 mg nivolumab IV over 60 minutes on day 1. Treatment repeats every 14 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease, complete response, or partial response receive 480 mg nivolumab IV over 60 minutes on day 1 of cycle 9. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 65 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Score [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 7
    1 | 4
    2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate for Participants Who Achieve a CR or PR [CT-based Response]
Description: The response rate for participants who achieve a CR or PR is defined as the percentage of participants who achieve a CR or PR assessed according to the revised Lugano Classification Response criteria. Complete response (CR): target nodes/nodal masses must regress to <=1.5 cm in longest transverse diameter (LDi). Partial response (PR): >= 50% decrease in sum of the product of the diameters (SPD) of up to 6 target measurable nodes and extranodal sites.
Time Frame: Up to 390 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 12
percentage of participants | 33.3 [12.3 to 63.7]

2. Secondary Outcome: Response Rate for Participants Who Achieve a CMR or PMR [PET-CT-based Response]
Description: The response rate for participants who achieve a CMR or PMR is defined as the percentage of participants who achieve a CMR or PMR assessed according to the revised Lugano Classification Response criteria. Complete metabolic response (CMR): Score 1, 2, or 3 with/without a residual mass using the Lugano 5-Point Scale (5-PS). Partial metabolic response (PMR): Score 4 or 5 with reduced update from baseline. The Lugano 5-PS is a scale used for initial staging and assessment of treatment response in Hodgkin lymphoma (HL) and certain types of non-Hodgkin lymphomas (NHL). The scale ranges from 1 to 5, where 1 is best and 5 is the worst. Each FDG-avid (or previously FDG-avid) lesion is rated independently: 1. no uptake or no residual uptake 2. slight uptake, but equal to or below blood pool 3. uptake above mediastinal, but below or equal to uptake in the liver 4. uptake slightly to moderately higher than liver 5. markedly increased uptake or any new lesion (on response evaluation)
Time Frame: Up to 390 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 12
percentage of participants | 33.3 [12.3 to 63.7]

3. Secondary Outcome: Duration of Response (DOR)
Description: The distribution of duration of response (CR or PR) will be estimated using the method of Kaplan-Meier. Complete response (CR): target nodes/nodal masses must regress to <=1.5 cm in longest transverse diameter (LDi). Partial response (PR): >= 50% decrease in sum of the product of the diameters (SPD) of up to 6 target measurable nodes and extranodal sites.
Time Frame: Up to 390 days
Population: Participants who achieved a response are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 4
months | 3.6 [1.9 to 6.9]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. In addition, the progression-free survival rate will be reported. progressive disease (PD): a Lugano score of 4 to 5 with increasing intensity compared to baseline or any interim scan and/or any new FDG-avid focus consistent with malignant lymphoma.The Lugano 5-PS is a scale used for initial staging and assessment of treatment response in Hodgkin lymphoma (HL) and certain types of non-Hodgkin lymphomas (NHL). The scale ranges from 1 to 5, where 1 is best and 5 is the worst. Each FDG-avid (or previously FDG-avid) lesion is rated independently: 1. no uptake or no residual uptake 2. slight uptake, but equal to or below blood pool 3. uptake above mediastinal, but below or equal to uptake in the liver 4. uptake slightly to moderately higher than liver 5. markedly increased uptake or any new lesion (on response evaluation)
Time Frame: The time from registration to relapse or death due to any cause, an average of 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 12
months | 1.9 [1.5 to 8.7]

5. Secondary Outcome: Overall Survival (OS)
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: The time from registration to death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 12
months | 7.9 [3.4 to 10.8]

6. Secondary Outcome: Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Events
Description: The number of participants who experienced at least one grade 3 or higher adverse events are summarized below.
Time Frame: Up to 390 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 12
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to 390 days
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 7/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=12)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Infections and infestations - Oth spec (Infections and infestations) | 2 (3)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=12)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (12)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (9)
Neutrophil count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (3)
Serum amylase increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT03075553/Prot_SAP_000.pdf